CLINICAL TRIAL: NCT00843284
Title: Assessing the Treatment of Patients With Neuropathic Pain Using LYRICA; A Non Interventional Post-marketing Study (NI-PMS)
Brief Title: Symptomatic Treatment Of Patients With Neuropathic Pain With LYRICA
Acronym: NI-PMS
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081139; ATLAS
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2009-04-16 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2009-10

CONDITIONS: Neuropathic Pain
Keywords: neuropathic, pain, pregabalin, Lyrica
MeSH Terms: conditions — Neuralgia; Pain | interventions — Pregabalin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with neuropathic pain
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Capsules, 150 - 600 mg/day, 2-3 times/day, 8 weeks

SUMMARY:
A Non-Interventional, Post-Marketing Surveillance (NI-PMS) study whose objectives were to assess the impact of pregabalin on subjects' pain, quality of sleep, and their general wellbeing, as well as the tolerance and safety of pregabalin in subjects with neuropathic pain.

DETAILED DESCRIPTION:
A non-interventional study of patients diagnosed with neuropathic pain administered pregabalin and followed up for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of neuropathic pain and inclusion according to the current Summary of Product Characteristics.

Exclusion Criteria:

* The patients were excluded according to the current Summary of Product Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuropathic pain
Sampling Method: Non-Probability Sample
Enrollment: 691 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081139&StudyName=Symptomatic%20Treatment%20Of%20Patients%20With%20Neuropathic%20Pain%20With%20LYRICA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 sites in Greece by investigators contracted by and under the direction of the sponsor. This study was performed by office-based physicians and in hospitals.
Pre-assignment Details: This study enrolled subjects with a confirmed diagnosis of neuropathic pain, according to the neuropathic pain diagnostic (DN4) Questionnaire, completed by the investigator at baseline
Groups:
- Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses): 275 subjects received pregabalin alone while 416 subjects received pregabalin in combination with another neuropathic pain medication.
Period: Overall Study
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Started | 691
Completed | 619
Not Completed | 72
Not completed — Adverse Event | 39
Not completed — Lack of Efficacy | 5
Not completed — Lost to Follow-up | 11
Not completed — Other | 10
Not completed — Withdrawal by Subject | 4
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Number analyzed (Participants) | 691
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (13.7)
Sex/Gender, Customized [Number; unit: participants]
  Female | 434
  Male | 254
  Unspecified | 3

OUTCOME MEASURES:

1. Secondary Outcome: Anxiety and Depression Symptoms
Description: The presence of anxiety and depression symptoms were measured, based on how often the subject felt a certain emotion over the past week. Q1:Have you felt calm and relaxed? Q2: Have you felt full of energy? Q3: Have you felt discouraged and sad? Final Visit = Week 8 or time of discontinuation.
Time Frame: Baseline, Final Visit (Week 8 or discontinuation)
Population: Full analysis set (FAS). Full analysis set was derived from the set of all enrolled subjects who were administered the study medication and had post baseline documentation of efficacy. Last observation carried forward method (LOCF) was used.
Measure: Number; unit: participants
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Number analyzed (Participants) | 668
participants
  Q1 at baseline: Always | 8
  Q1 at baseline: Most of the time | 14
  Q1 at baseline: Fairly often | 57
  Q1 at baseline: Sometimes | 199
  Q1 at baseline: Rarely | 186
  Q1 at baseline: Never | 183
  Q1 at baseline: Missing | 0
  Q1 at baseline: Not done | 21
  Q1 at final visit: Always | 27
  Q1 at final visit: Most of the time | 152
  Q1 at final visit: Fairly often | 168
  Q1 at final visit: Sometimes | 176
  Q1 at final visit: Rarely | 72
  Q1 at final visit: Never | 37
  Q1 at final visit: Missing | 1
  Q1 at final visit: Not done | 35
  Q2 at baseline: Always | 5
  Q2 at baseline: Most of the time | 15
  Q2 at baseline: Fairly often | 62
  Q2 at baseline: Sometimes | 150
  Q2 at baseline: Rarely | 196
  Q2 at baseline: Never | 219
  Q2 at baseline: Missing | 0
  Q2 at baseline: Not done | 21
  Q2 at final visit: Always | 21
  Q2 at final visit: Most of the time | 108
  Q2 at final visit: Fairly often | 168
  Q2 at final visit: Sometimes | 174
  Q2 at final visit: Rarely | 102
  Q2 at final visit: Never | 59
  Q2 at final visit: Missing | 1
  Q2 at final visit: Not done | 35
  Q3 at baseline: Always | 48
  Q3 at baseline: Most of the time | 167
  Q3 at baseline: Fairly often | 190
  Q3 at baseline: Sometimes | 143
  Q3 at baseline: Rarely | 59
  Q3 at baseline: Never | 40
  Q3 at baseline: Missing | 0
  Q3 at baseline: Not done | 21
  Q3 at final visit: Always | 7
  Q3 final visit: Most of the time | 37
  Q3 at final visit: Fairly often | 73
  Q3 at final visit: Sometimes | 179
  Q3 at final visit: Rarely | 161
  Q3 at final visit: Never | 175
  Q3 at final visit: Missing | 1
  Q3 at final visit: Not done | 35

2. Primary Outcome: Daily Average Pain Scores
Description: Change is observed value at final visit (Week 8 or discontinuation) minus baseline value. Daily average pain score is measured using a 10-point Likert scale where 0 = no pain to 10 = pain as bad as you can imagine.
Time Frame: Baseline, Final Visit (Week 8 or discontinuation)
Population: Full analysis set (FAS). Full analysis set was derived from the set of all enrolled subjects who were administered the study medication and had post baseline documentation of efficacy. Last observation carried forward (LOCF) method was used.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Number analyzed (Participants) | 668
scores on scale
  Baseline | 7.61 (1.69)
  Final visit (Week 8 or discontinuation) | 3.46 (2.11)
  Change from baseline | -4.16 (2.52)
Statistical Analysis 1: Comparison: Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses); Change from Baseline; observational study; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test; Mean Difference (Net) = -4.16, 95% CI [-4.35 to -3.97], Standard Deviation 2.52

3. Primary Outcome: Pain Related Sleep Interference
Description: Change is observed value at final visit (Week 8 or discontinuation) minus baseline value. Pain related sleep interference is measured by a 10-point Likert scale where 0 = does not interfere with sleep, and 10 = completely interferes with sleep
Time Frame: Baseline, Final Visit (Week 8 or discontinuation)
Population: Full analysis set (FAS) was derived from the set of all enrolled subjects who were administered the study medication and had post baseline documentation of efficacy. Last observation carried forward (LOCF) method was used.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Number analyzed (Participants) | 668
scores on a scale
  Baseline | 6.28 (2.59)
  Final visit (Week 8 or discontinuation) | 2.27 (2.19)
  Change from baseline | -4.02 (2.90)
Statistical Analysis 1: Comparison: Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses); Change from baseline; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; One sample t-test; Mean Difference (Net) = -4.02, 95% CI [-4.24 to -3.80], Standard Deviation 2.90

4. Secondary Outcome: Clinician Global Improvement of Change (CGIC) at Final Visit (Week 8 or Discontinuation)
Description: Clinician Global Improvement of Change (CGIC) indicates the change of the severity of the condition from baseline, graded from "very much improved" to "very much worse".
Time Frame: Final Visit (Week 8 or discontinuation)
Population: Full analysis set (FAS). Full analysis set was derived from the set of all enrolled subjects who were administered the study medication and had post baseline documentation of efficacy. Last observation carried forward (LOCF) method was used. Three subjects were not included in the analysis due to incomplete case report forms.
Measure: Number; unit: participants
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Number analyzed (Participants) | 665
participants
  Not assessed | 0
  Very much improved | 160
  Much improved | 292
  Minimally improved | 171
  No change | 39
  Minimally worse | 1
  Much worse | 2
  Very much worse | 0
  Not done | 0

5. Secondary Outcome: Patient Global Improvement of Change (PGIC) at Final Visit (Week 8 or Discontinuation)
Description: Patient Global Improvement of Change (PGIC) indicates the change of severity of conditions from baseline, graded from "very much improved" to "very much worse".
Time Frame: Final Visit (Week 8 or discontinuation)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Number analyzed (Participants) | 666
participants
  Not assessed | 0
  Very much improved | 175
  Much improved | 245
  Minimally improved | 193
  No change | 44
  Minimally worse | 7
  Much worse | 2
  Very much worse | 0
  Not done | 0

ADVERSE EVENTS:
Arm/Group | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Serious Adverse Events (participants affected / at risk) | 7
Other Adverse Events (participants affected / at risk) | 151
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Cardiopulmonary failure (Cardiac disorders) | 1/691
Abdominal pain (Gastrointestinal disorders) | 1/691
Nausea (Gastrointestinal disorders) | 1/691
Asthenia (General disorders) | 1/691
Death (General disorders) | 3/691
Fatigue (General disorders) | 1/691
Tremor (Nervous system disorders) | 1/691
Dysphoria (Psychiatric disorders) | 1/691
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/691
Walking disability (Social circumstances) | 1/691
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pregabalin (150 mg to 600 mg Per Day in 2 to 3 Divided Doses)
Dizziness (Nervous system disorders) | 133/691
Somnolence (Surgical and medical procedures) | 67/691

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.